CLINICAL TRIAL: NCT02802852
Title: Proteomics and Stem Cell Therapy as a New Vascularization Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, George Havelka MD MS RPVI, Assistant Professor of Surgery, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1244
Record Dates: First submitted 2016-04-21; First posted 2016-06-16 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calf Compression, Filgrastim injection (Experimental): All patients enrolled in the study will undergo pneumatic calf compression though use of the Art Assist device as well as stem cell mobilization through administration of Filgrastim 10 mcg/kg subcutaneously, every 3rd day for 30 days.
  Interventions: Device: Pneumatic calf compression; Drug: Filgrastim

INTERVENTIONS:
Device: Pneumatic calf compression — Application of a pneumatic calf compression device for two hours per day, every day for 30 days.
  Other Names: Art Assist Device
Drug: Filgrastim — Administration of Filgrastim 10 mcg/kg every 3rd day for 30 days
  Other Names: Neupogen

SUMMARY:
Neovascularization (NV) is the innate capability to enlarge collateral arteries ("arteriogenesis"), and to stimulate growth of new capillaries, arterioles and venules at the tissue level ("angiogenesis"). Patients with Chronic Limb-threatening Ischemia (CLI) present with forefoot rest-pain, ulceration and/or gangrene. They require risky and costly revascularization operations to avoid amputation. The investigators hypothesize that their inadequate NV can be modulated to restore this capability. By correcting impediments to NV in an out-patient setting, the investigators expect to facilitate CLI management.

While the following impediments to NV are complex, the solution is not. Arteriogenesis necessitates endothelial cell activation in small collaterals as blood is offloaded away from the occluded artery. Shear stress provides this stimulus, but is attenuated caudal to multi-level arterial occlusive disease. The "arteriogenesis switch" is not turned on. Furthermore, the lack of nutritive oxygenated blood inflow and the accumulation of toxic metabolic by-products are adverse to synthetic pathways in the ischemic tissue. Additionally, protein "distress" signals cannot be effectively disseminated by the ischemic tissue, and the reparative progenitor cells they are supposed to mobilize cannot effectively home back to the ischemic tissue to orchestrate NV. The CLI patient is especially disadvantaged by having diminished function and number of circulating progenitor cells (CPC). Lastly these elderly, often diabetic, patients are less able to fend off infection.

An FDA approved external programmed pneumatic compression device (PPCD) was used to restore the shear stress stimulus required for arteriogenesis. It also enhances oxygenated nutritive arterial inflow, clears waste products of metabolism (increased venous and lymphatic outflow), and helps distress proteins reach the central circulation and mobilized progenitor cells to return to the ischemic tissue. We corrected the progenitor cell and immunologic impairment with granulocyte colony stimulating factor (G-CSF), FDA approved for stem cell mobilization and immunological boost in the setting of cancer chemotherapy. The preliminary data show clinical, angiographic, hemodynamic and biochemical evidence for enhanced NV. The purpose for this study is to enroll 25 patients to reproduce the biochemical data to support a large scale clinical trial.

DETAILED DESCRIPTION:
Twenty-five CLI patients with ischemic forefoot rest pain, non-healing forefoot ulceration, or dry forefoot gangrene will be recruited. They will have already undergone standard of care evaluation, including hemodynamic testing and duplex ultrasound delineation of the arterial anatomy in the Non-invasive Vascular Laboratory. Those with tibial artery occlusive disease, with normal or corrected proximal aorto-ilio-femoral arterial anatomy, will be given the option of enrollment in lieu of surgery or catheter revascularization.

The standard vascular assessment data will be reviewed: History and Physical (H&P) examination, vascular laboratory hemodynamic data (arterial duplex imaging, ankle and toe pressures), and blood tests (complete blood cell count, metabolic and lipid panel, hemoglobin A1C if diabetic). Carotid duplex scan, chest X-Ray, electrocardiogram, chemical cardiac stress test, and echocardiogram will be reviewed if available. While angiography by magnetic resonance imaging (MRI), computed tomography(CT) or catheter may be available, they are not required. Data obtained from in-clinic use of LUNA fluorescence angiography may also be collected, but is not necessary. To emphasize, all ultrasound, x-ray, CT, MRI and LUNA fluorescence data may be collected since imaging is the standard of care for patients being evaluated for peripheral vascular disease, but no specific imaging is required and no imaging is being studied as part of this protocol.

PPCD use will continue until the presenting symptoms resolve or traditional revascularization becomes necessary to achieve limb salvage. Each patient serves as his/her own control. Three "pairs" of blood specimens will be analyzed per patient. A "pair" includes phlebotomy prior to and immediately after two hours of PPCD. The first pair is obtained on enrollment in the study. The second pair will be done 2 weeks later 18-24 hours after the last dose of G-CSF. The third pair will be done 30 days into the study, 18-24 hours after the last dose of G-CSF. The patient will return for standard of care clinical evaluation, with repeat hemodynamic testing, 6 months after the 30 day clinic evaluation.

Case Report Forms (CRFs) will be prepared for each subject. Progression of ischemic symptoms will result in discontinuation of participation in the trial and immediate standard of care treatment, including imaging studies and revascularization, if indicated. Otherwise the status of the presenting forefoot symptoms (ischemic rest pain, ischemic ulcers, and gangrene) will be documented at Day 1, Day 14, and Day 30. Ischemic rest pain will be scored (1 to 10 scale). Pain free walking distance will be measured. Forefoot ischemic lesions will be photographed and dimensions recorded on enrollment.

Baseline visit (Outpatient Care Center):

1. Patents will undergo standard of care H&P examination.
2. Upon verification that the patient is eligible (based on the inclusion/exclusion criteria), an informed consent form will be explained to the patient to better explain the study and ask for authorization to participate.

Baseline visit (Non-invasive Vascular Ultrasound Laboratory):

1. Other standard of care tests will include: duplex ultrasound (DUS), ankle and toe pressures, if not yet completed prior to the clinic visit.

Day1 (Clinical Resource Center, University of Illinois at Chicago): The following procedures will be done in this order:

1. Initial blood draw (20 ml)
2. Patients then will wear the PPCD in seated position (2-hour session).
3. After the 2-hour use of the PPCD, another blood draw will be done (20 ml).
4. Each patient will be given a Neupogen shot (10 mcg/kg) subcutaneously
5. Patient will be given ample time to fill out the quality of life (QOL) questionnaires (SF36, EQ5D, VascQoL-6) and a study coordinator will be available at this time to assist the patient. Each questionnaire will take about 10 minutes to fill out.
6. Blood samples will be sent to the Dr. Bartholomew, MD Lab for analysis.

Days 4, 7, 10, and 13 (at Home or in clinic): The following procedures will be done:

1. Nurse or PI will administer a Neupogen shot (10 mcg/kg) subcutaneously, every 3rd day, for a total of 10 Neupogen shots. Patient will continue use of the PPCD every day, at least 3 hours a day, till symptoms are resolved.

Day14 (Clinical Resource Center, University of Illinois at Chicago): The following procedures will be done in this order:

1. Initial blood drawing (20 ml), 18-24 hours after the 5th shot of Neupogen. Blood samples will be sent to Dr. Bartholomew Lab for biochemical analysis.
2. Patients will then wear PPCD for 2 hours in seated position.
3. Just prior to the end of the 2-hour use of the PPCD, another blood draw will be done (20 ml).
4. Patient will return the empty vials of Neupogen.
5. Patient will be given ample time to fill out the quality of life (QOL) questionnaires (SF36, EQ5D, VascQoL-6) and a study coordinator will be available at this time to assist the patient. Each questionnaire will take about 10 minutes to fill out.

Day30 (Clinical Resource Center, University of Illinois at Chicago): The following procedures will be done in this order:

1. Initial blood drawing (20 ml), 18-24 hours after the 10th shot of Neupogen. Blood samples will be sent to Dr. Bartholomew Lab for biochemical analysis.
2. Patients will then wear PPCD for 2 hours in seated position.
3. Just prior to the end of the 2-hour use of the PPCD, another blood draw will be done (20 ml).
4. Patient will be given ample time to fill out the quality of life (QOL) questionnaires (SF36, EQ5D, VascQoL-6) and a study coordinator will be available at this time to assist the patient. Each questionnaire will take about 10 minutes to fill out.
5. Patient will return the empty vials of Neupogen.

Monthly Follow-up (Clinical Resource Center, University of Illinois at Chicago):

1. After the completion of the initial 30 day treatment period, the patient will follow-up in clinic at 1 month intervals for ongoing clinical assessment. The patient will continue using the device alone daily until wounds are healed and forefoot rest pain has resolved.
2. At 6 month visit, the patient will fill out QOL questionnaires. Each patient will be followed for a total of 6 months. Repeat hemodynamic testing will occur in our Intersocietal Accreditation Commission certified non-invasive ultrasound laboratory at the 6 month visit.

Unscheduled visits and early termination:

1. Enrolled subjects will be given the contact information for the principal investigator so that they can have access to the study organizers should any questions or concerns arise at home in-between clinic visits. Patients wishing to terminate their enrollment in the study can contact the principal investigator in the same manner.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 35 and 85.
2. Chronic limb ischemia Fontaine Class III (ischemic forefoot rest pain) and Class IV (non-healing ischemic ulcers, gangrene) with confirmatory non-invasive vascular testing.
3. English or Spanish speaking patients

Exclusion Criteria:

1. Acute limb ischemia requiring emergency treatment.
2. Non-salvageable foot (e.g. extensive gangrene, advanced infection, rigor mortis, knee/hip flexion contracture, post-stroke paralysis, and hemiparesis).
3. Untreated hypercoagulability disorder, sickle cell anemia, myeloproliferative disorder.
4. Dialysis, and/or sustained elevated Creatinine >3.6 mg/dl.
5. Severe dementia; bed-ridden; non-compliance; unlikely to follow-up; unreliable.
6. Intolerance of PPCD compression
7. Morbid obesity (Body Mass Index > 34)
8. Severe venous insufficiency causing venous stasis ulceration and dermatitis.
9. Uncorrected significant aorto-iliac, common femoral, and profunda femoral arterial disease
10. Ulceration precluding PPCD placement.
11. Active cancer.
12. Allergy to Neupogen.
13. Uncorrected symptomatic coronary artery disease
14. History of lymphoma or leukemia

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Hepatocyte Growth Factor | Change between 1 day, 14 days, and 30 days
Insulin Growth Factor | Change between 1 day, 14 days, and 30 days
Vascular Endothelial Growth Factor A | Change between 1 day, 14 days, and 30 days
Vascular Endothelial Growth Factor B | Change between 1 day, 14 days, and 30 days
Vascular Endothelial Growth Factor C | Change between 1 day, 14 days, and 30 days
Vascular Endothelial Growth Factor 165b | Change between 1 day, 14 days, and 30 days
Matrix Metalloproteinase 9 | Change between 1 day, 14 days, and 30 days
Tissue Necrosis Factor alpha | Change between 1 day, 14 days, and 30 days
Placental Growth Factor | Change between 1 day, 14 days, and 30 days
Platelet Derived Growth Factor AA | Change between 1 day, 14 days, and 30 days
Platelet Derived Growth Factor BB | Change between 1 day, 14 days, and 30 days
Angiopoietin | Change between 1 day, 14 days, and 30 days
Tissue Growth Factor beta | Change between 1 day, 14 days, and 30 days
Plasmin | Change between 1 day, 14 days, and 30 days
Fibrin Degradation Products | Change between 1 day, 14 days, and 30 days
Interleukin 6 | Change between 1 day, 14 days, and 30 days
Interleukin 8 | Change between 1 day, 14 days, and 30 days
CD 34+ Cytometry | Change between 1 day, 14 days, and 30 days
Vascular Endothelial Growth Factor Receptor 2+ Cytometry | Change between 1 day, 14 days, and 30 days
CD 14+ Cytometry | Change between 1 day, 14 days, and 30 days
CD 31+ Cytometry | Change between 1 day, 14 days, and 30 days
Serum Nitrate | Change between 1 day, 14 days, and 30 days

SECONDARY OUTCOMES:
Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) | 14 days, 30 days, 6 months
  The generic Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) self-administered questionnaire will be completed with assistance from the PI and co-investigators at the initial visit, on Days 14 and 30 as well as at 6 months. The SF-36 covers physical and social function, and role limitations due to physical and emotional problems, mental health, energy and vitality, pain, and general health.
Vascular Quality of Life Questionnaire | 14 days, 30 days, 6 months
  The Vascular Quality of Life Questionnaire (VascuQol) self-administered questionnaire will be completed with assistance from the PI and co-investigators at the initial visit, on Days 14 and 30 as well as at 6 months. The VascuQol is a peripheral artery disease score of activity, symptom, pain, emotion, and social function.
EuroQol-5D | 14 days, 30 days, 6 months
  The EuroQol-5D self-administered questionnaire will be completed with assistance from the PI and co-investigators at the initial visit, on Days 14 and 30 as well as at 6 months. The EuroQol-5D covers mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: George E Havelka, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eton D, Yu H. Enhanced cell therapy strategy to treat chronic limb-threatening ischemia. J Vasc Surg. 2010 Jul;52(1):199-204. doi: 10.1016/j.jvs.2009.12.048. Epub 2010 Mar 28. PMID 20347552
- [Background] Rauscher FM, Goldschmidt-Clermont PJ, Davis BH, Wang T, Gregg D, Ramaswami P, Pippen AM, Annex BH, Dong C, Taylor DA. Aging, progenitor cell exhaustion, and atherosclerosis. Circulation. 2003 Jul 29;108(4):457-63. doi: 10.1161/01.CIR.0000082924.75945.48. Epub 2003 Jul 14. PMID 12860902
- [Background] Fadini GP, Avogaro A. Autologous transplantation of granulocyte colony-stimulating factor- mobilized peripheral blood mononuclear cells improves critical limb ischemia in diabetes. Diabetes Care. 2006 Feb;29(2):478-9; author reply 479-80. doi: 10.2337/diacare.29.02.06.dc05-1770. No abstract available. PMID 16482702
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Derived] Eton D, Zhou G, He TC, Bartholomew A, Patil R. Filgrastim, fibrinolysis, and neovascularization. J Tissue Eng Regen Med. 2022 May;16(5):496-510. doi: 10.1002/term.3284. Epub 2022 Feb 17. PMID 35175691